CLINICAL TRIAL: NCT01600170
Title: Statin Modulation of Monocyte/Macrophage Activation for HAND Treatment
Brief Title: Downmodulating Monocyte Activation for HIV-1 Associated Neurocognitive Disorders (HAND)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Protocol # 815512
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: HIV Dementia
Keywords: HIV; monocytes; CD16+; statins; mcp1; inflammation
MeSH Terms: conditions — AIDS Dementia Complex; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): Participants were given atorvastatin for 12 weeks at various doses based on their specific HAART treatment.
  Interventions: Drug: Atorvastatin (generic Lipitor)
- Placebo (Placebo Comparator): Participants were given Placebo tablets for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin (generic Lipitor) — Atorvastatin is an FDA approved prescription drug which is frequently used to lower cholesterol levels.It is available in the form of tablets ranging in dose from 10-80mg.
  Arms: Atorvastatin
Drug: placebo — A substance containing no medication and prescribed or given to reinforce a patient's expectation to get well.
  Arms: Placebo

SUMMARY:
HIV associated neurological disorders (HAND), are a major problem even in ART treated people. HAND results from chronic inflammation which is largely attributed to expansion and activation of monocytes. These activated monocytes, some of which also carry virus to the brain, invade the CNS and release cytokines / chemokines resulting in further recruitment of monocytes, as well as release viral proteins which injure neurons and cause activation of other brain cells. Persistent monocyte/macrophage activation is thus a potential critical target for adjunctive therapy to treat or prevent HAND. The investigators therefore propose to study the effects of a statin drug (Atorvastatin), which has anti-inflammatory functions, on the monocyte activation status in ART treated HIV+ individuals.

The investigators objectives are based on the hypothesis that Atorvastatin treatment will reduce the inflammatory and activated phenotype and function of monocytes which have been linked to HIV associated neuropathogenesis and occur in HIV infected subjects despite ART. In this study the investigators propose to

1) define the effect of Atorvastatin on monocyte activation in HIV infected / ART treated subjects in a double blind, placebo controlled crossover study

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HIV-1 infected individuals on HAART (with no change in treatment within 4 weeks of study entry) and willing to continue therapy for the duration of the study.
2. HIV viral load less than 200 copies/ml for more than 6 months at time of screening.
3. Nadir CD4 count less than 350 and current CD4 counts greater than 100 cells/ul.
4. Hs-CRP levels above 2mg/L.
5. Willingness to use a method of contraception during the study period.
6. Willingness to comply with study evaluations for LP sub-study.
7. Karnofsky performance score of 80 or higher.
8. If female, willing to undergo pregnancy testing on a monthly basis and not breastfeeding.
9. Hemoglobin greater than or equal to 9.0 g/dL for female and 10.0 g/dL for male subjects.
10. men and women 18 years or older.

Exclusion Criteria:

1. Concomitant use of fibric acid derivatives or other lipid lowering agents including patients on statins and Ezetimibe.
2. Use of any anti-inflammatory drugs (OTC or prescription) on a daily basis.
3. Pregnancy or breastfeeding
4. Active drug use or alcohol abuse/dependence which in the opinion of researchers will interfere with the patients' ability to participate in the study.
5. Allergy or hypersensitivity to Atorvastatin or any of its components.
6. History of myositis or rhabdomyolysis with use of any statins.
7. Patients who are on concurrent immunomodulatory agents, including systemic corticosteroids (nasal or inhaled) will be ineligible for 3 months after completion of therapy with the agent.
8. History of inflammatory muscle disease such a poly or dermatomyositis.
9. Serious intercurrent illness requiring systemic treatment and/or hospitalization within 30 days of entry.
10. Evidence of active opportunistic infections requiring treatment or neoplasms that require chemotherapy during study period.
11. CPK greater than 3 times the ULN.
12. Known active liver disease or AST/ALT greater than 3 times the ULN.
13. Renal insufficiency, indicated by serum creatinine greater than 2mg/dL.
14. Absolute neutrophil counts less than 1000/ul; hemoglobin less than 10g/dL for males and less than 9g/dL for females; platelet counts less than 100,000/mm3.
15. Documented HCV infection.
16. NYHA class III or IV congestive heart failure.
17. Active IV drug use within 1 year prior to entry.
18. For LP sub-study, allergy to Lidocaine.
19. Coronary artery disease or equivalent including Diabetes mellitus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Collman, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic HIV infected individuals on HAART (with no changes in treatment within 4 weeks of study entry), were recruited using the Penn CFAR Clinical Core database. Subject were consented by the study nurse coordinating the project. Of 46 screened subjects, 11 fulfilled the inclusion criteria and were enrolled in the study.
Pre-assignment Details: Participants that met the inclusion criteria were randomly assigned to 12weeks of atorvastatin (or placebo) in the first period followed by a 4week washout and then in the second period on placebo (or atorvastatin) for 12 weeks followed by washout (4weeks). Therefore each subject served as their own control.
Groups:
- Atorvastatin, Then Placebo: Participants were assigned atorvastatin at different conc. (20, 40 or 60mg / day) based on HAART for 12 wks. After a washout period of 4 weeks participants received placebo tablets (matching atorvastatin), for 12 weeks followed by another washout period of 4 weeks.
- Placebo, Then Atorvastatin: Participants were assigned placebo tablets for 12 wks. After a washout period of 4 weeks participants received atorvastatin tablets at different conc.(20, 40 or 60mg / day) based on HAART, for 12 weeks followed by another washout period of 4 weeks.
Period: Period 1
Arm/Group | Atorvastatin, Then Placebo | Placebo, Then Atorvastatin
Started | 6 (Participants were assigned atorvastatin for 12 wks followed by a washout and then placebo.) | 5 (Participants were assigned placebo for 12 wks followed by a washout and then atorvastatin.)
Completed | 6 | 5
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Atorvastatin, Then Placebo | Placebo, Then Atorvastatin
Started | 6 (These 6 were on atorvastatin in period 1 and on placebo in Period 2.) | 5 (These 5 were on placebo in Period 1 and on Atorvastatin in Period 2.)
Completed | 5 (One subject moved away from the area due to job responsibilities and dropped out of study.) | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin Then Placebo: Participants were given Atorvastatin followed by a washout period then placebo.
  1. Subjects on PI based HAART regimen were administered atorvastatin at 10mg/day X 2weeks and then 20mg/day for 10 weeks.
  2. Subjects on non-PI / non-NNRTI based HAART regimen were administered 20mg/day X 2weeks and then 40mg/day X 10weeks.
  3. Subjects on NNRTI based HAART regimen were administered 40mg/day X 2weeks and then 80mg/day X 10weeks.
- Placebo Then Atorvastatin: Participants were administered Placebo tablets followed by a washout period and then Atorvastatin.
  1. Subjects on PI based HAART regimen were administered atorvastatin at 10mg/day X 2weeks and then 20mg/day for 10 weeks.
  2. Subjects on non-PI / non-NNRTI based HAART regimen were administered 20mg/day X 2weeks and then 40mg/day X 10weeks.
  3. Subjects on NNRTI based HAART regimen were administered 40mg/day X 2weeks and then 80mg/day X 10weeks.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin Then Placebo | Placebo Then Atorvastatin | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.8) | 47.9 (12.0) | 45.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 0 | 1 | 1
  African American | 6 | 4 | 10
  Ethnicity: Non Hispanic / Latino | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 in Percentage of Blood Monocytes Expressing Surface Marker CD16 at 12 Weeks, as a Result of Treatment.
Description: Whole blood drawn from participants were stained with fluorochrome tagged antibodies to the surface markers. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the change in percentage of monocytes expressing the specific marker (CD16) at 12 wk versus 0wk within each Period.
  Data is shown as fold change over 12 weeks, in percent positive monocytes expressing surface markers.
  Change in primary outcome measures in each treatment arm is expressed as fold change (at week 12 versus week 0). For eg. outcome measure CD14+CD16+ in atorvastatin arm shows a mean value of 1.14. This means at 12 weeks there is an increase of 0.14 fold in the percent monocyte population expressing CD14+CD16+ marker, versus 0 week. Similarly in the placebo group. If fold change in atorvastatin group is smaller than in placebo group, then the treatment had no effect.
Time Frame: Week 0 and week 12
Population: Subjects received Atorvastatin or placebo for 12wks followed by 4wk washout period then switched treatment for 12 wks followed again by a washout period. The same 11 subjects were analyzed in each group.
Measure: Mean (95% Confidence Interval); unit: Fold change
Groups:
- Atorvastatin: Participants were given Atorvastatin depending on their HAART
  1. Subjects on PI based HAART regimen were administered atorvastatin at 10mg/day X 2weeks and then 20mg/day for 10 weeks.
  2. Subjects on non-PI / non-NNRTI based HAART regimen were administered 20mg/day X 2weeks and then 40mg/day X 10weeks.
  3. Subjects on NNRTI based HAART regimen were administered 40mg/day X 2weeks and then 80mg/day X 10weeks.
- Placebo: Participants were administered Placebo tablets for 12 weeks.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold change | 1.14 [0.73 to 1.77] | 1.51 [0.88 to 2.59]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Analysis focused on a comparison of change in response over 12 wks for each treatment under a 2x2 crossover design. Mixed effects model was used to estimate within subject treatment differences, trends over time & at each wk(0,2,6,12). Log-transformations were applied to meet normality assumption & models adjusted for period & sequence effects. Primary outcomes were pre-specified to use p<0.01 for statistical significance. All other analyses used p<0.05 after adjustment for multiple comparisons; Test type: Superiority; p = 0.39, Mixed Models Analysis — The threshold for statistical significance was p = 0.01

2. Primary Outcome: Change From Baseline Within Each Period in Levels of Plasma Inflammatory Marker MCP-1 in Chronic HIV+/ HAART+ Subjects Over 12 Weeks.
Description: Monocyte specific inflammatory soluble factor MCP-1 was measured by Luminex in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following treatment (atorvastatin or placebo).
  Data is shown as fold change in concentration of MCP-1 over 12wks within each treatment period.
Time Frame: Week 0 and week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold change
Groups:
- Atorvastatin: Participants were given Atorvastatin based on their HAART
  1. Subjects on PI based HAART regimen were administered atorvastatin at 10mg/day X 2weeks and then 20mg/day for 10 weeks.
  2. Subjects on non-PI / non-NNRTI based HAART regimen were administered 20mg/day X 2weeks and then 40mg/day X 10weeks.
  3. Subjects on NNRTI based HAART regimen were administered 40mg/day X 2weeks and then 80mg/day X 10weeks.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold change | 0.96 [0.82 to 1.13] | 0.87 [0.67 to 1.12]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.45, Mixed Models Analysis — Threshold of statistical significance was p=0.01

3. Primary Outcome: Change From Week 0 in Percentage of Blood Monocytes Expressing Surface Marker CD163 at 12 Weeks, as a Result of Treatment.
Description: Whole blood drawn from participants were stained with fluorochrome tagged antibodies to the surface marker CD163. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the change in percentage of monocytes expressing the specific marker (CD163) at 12 wk versus 0wk within each Period.
  Data in each treatment arm is shown as 'mean difference' at 12 weeks versus 0 week, in percent positive monocytes expressing surface marker CD163.
  Data is expressed as the difference of the mean values at week 12 and week 0. The negative values mean that the mean values at 12 week were lower than the mean values at 0 week.
Time Frame: week 0 and week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of monocytes
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Percentage of monocytes | -0.06 [-9.17 to 9.05] | -5.14 [-11.94 to 1.65]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.80, Mixed Models Analysis — The threshold for statistical significance was p = 0.01

4. Primary Outcome: Change From Week 0 in Percentage of Blood Monocytes Expressing Surface Marker CCR2 at 12 Weeks, as a Result of Treatment.
Description: Whole blood drawn from participants were stained with fluorochrome tagged antibodies to the surface marker CCR2. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the change in percentage of monocytes expressing the specific marker (CCR2) at 12 wk versus 0wk within each Period.
  Data in each treatment arm is shown as fold change over 12 weeks, in percent positive monocytes expressing surface marker CCR2.
Time Frame: week 0 and week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change | 1.60 [0.80 to 3.21] | 0.78 [0.52 to 1.18]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Mixed Models Analysis — The threshold of statistical significance was p=0.01

5. Primary Outcome: Change From Baseline Within Each Period in Levels of Plasma Inflammatory Marker sCD14 in Chronic HIV+/ HAART+ Subjects Over 12 Weeks.
Description: Monocyte specific inflammatory soluble factor sCD14 was measured by ELISA in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following treatment (atorvastatin or placebo).
  Data is shown as fold change in concentration of sCD14 over 12wks within each treatment period.
Time Frame: 0 week and 12 week
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change | 0.95 [0.80 to 1.12] | 1.04 [0.94 to 1.16]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.15, Mixed Models Analysis — The threshold of statistical significance was p=0.01

6. Secondary Outcome: Change From Week 0 to Week 12 in Percentage of Blood Monocytes Expressing Surface Marker Tissue Factor (TF), Following Treatment.
Description: Whole blood drawn from participants were stained with fluorochrome tagged antibodies to the surface marker TF. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the change in percentage of monocytes expressing the specific marker TF at 12 wk versus 0wk within each Period.
  Data are expressed as fold change.
Time Frame: 0 week and 12 week
Population: Subjects were assigned to Atorvastatin or placebo for 12wks followed by 4wk washout period then subjects switched treatment for 12 wks followed again by a washout period. The same 11 subjects were analyzed in each group.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold change | 1.18 [0.57 to 2.42] | 1.52 [0.75 to 3.09]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Analysis focused on a comparison of change in response over 12 wks for each treatment under a 2x2 crossover design. Mixed effects model was used to estimate within subject treatment differences, trends over time & at each wk(0,2,6,12). Log-transformations were applied to meet normality assumption & models adjusted for period & sequence effects. Secondary outcome analyses used p<0.05 for statistical significance after adjustment for multiple comparisons; Test type: Superiority; p = 0.63, Mixed Models Analysis — The threshold for statistical significance was p = 0.05

7. Secondary Outcome: Change From 0 Week in Levels of Plasma Inflammatory Marker hsCRP in Chronic HIV+/ HAART+ Subjects Over 12 Weeks, Following Treatment.
Description: Monocyte specific inflammatory soluble factor hsCRP was measured by Quest in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following treatment (atorvastatin or placebo).
  Data shown as fold change at week 12 versus week 0.
Time Frame: 0 week and 12 week
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold change | 0.94 [0.61 to 1.44] | 1.70 [0.85 to 3.39]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.035, Mixed Models Analysis — Threshold for statistical significance was p = 0.05

8. Secondary Outcome: Change From Week 0 to Week 12 in Percentage of Blood Monocytes Expressing Surface Marker CD38, Following Treatment.
Description: Whole blood drawn from participants were stained with fluorochrome tagged antibodies to the surface marker CD38. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the change in percentage of monocytes expressing the specific marker CD38 at 12 wk versus 0wk within each Period.
  Data are expressed as fold change at 12 week versus week 0.
Time Frame: 0 week and 12 week
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change | 0.98 [0.86 to 1.12] | 1.04 [0.86 to 1.27]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.62, Mixed Models Analysis — The threshold of statistical significance was p = 0.05

9. Secondary Outcome: Change From Week 0 in Plasma sCD163 Levels, at Week 12 Following Treatment.
Description: Monocyte specific inflammatory soluble factor sCD163 was measured by ELISA in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following treatment (atorvastatin or placebo).
  Data are expressed as fold change at 12 week versus week 0.
Time Frame: 0 week and 12 week
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change | 1.08 [0.97 to 1.2] | 1.02 [0.85 to 1.22]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.99, Mixed Models Analysis — The threshold of statistical significance was p = 0.05

ADVERSE EVENTS:
Time Frame: Participants were observed for the duration of the study enrollment period, i.e. 36 weeks.
Description: Participants were routinely assessed for any adverse events with regular laboratory testing, and study Investigator and study nurse assessment.
Groups:
- Atorvastatin: Participants were given Atorvastatin for 12 weeks based on HAART
  1. Subjects on PI based HAART regimen were administered atorvastatin at 10mg/day X 2weeks and then 20mg/day for 10 weeks.
  2. Subjects on non-PI / non-NNRTI based HAART regimen were administered 20mg/day X 2weeks and then 40mg/day X 10weeks.
  3. Subjects on NNRTI based HAART regimen were administered 40mg/day X 2weeks and then 80mg/day X 10weeks.
Arm/Group | Atorvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
This study had a very small sample size of 11 subjects and did not reach target recruitment (30 subjects) due to stringent study Inclusion criteria. Therefore due to lack of power the data is largely inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT01600170/Prot_SAP_000.pdf